CLINICAL TRIAL: NCT01497847
Title: Post-Infectious Irritable Bowel Syndrome (PI-IBS)
Acronym: PI-IBS
Status: Completed | Type: Observational
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Guy Boeckxstaens, Principal Investigator, KU Leuven
Other Study IDs: S51501
Record Dates: First submitted 2011-12-16; First posted 2011-12-23 (Estimated); Last update posted 2013-04-26 (Estimated); Status verified 2013-04

CONDITIONS: Irritable Bowel Syndrome With Diarrhea
Keywords: Post-Infectious Irritable Bowel Syndrome; PI-IBS

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, blood plasma, feces, rectal biopsy
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- travelers to tropical destinations

SUMMARY:
Purpose:

* identification of factors predisposing for Post-Infectious Irritable Bowel Syndrome (PI-IBS) development after an episode of traveler's diarrhea
* identification of systemic (serum) and local (biopsy) changes in infectious and immunological activity during infection and correlation with Irritable Bowel Syndrome (IBS) symptoms, persisting after traveler's diarrhea

Design:

* 4 study visits: before traveling, 2 weeks after traveling, 6 months after traveling, 12 months after traveling
* at each study visit following investigations: blood collection, stool collection, questionnaires, rectal biopsy

ELIGIBILITY:
Inclusion Criteria:

* traveling to South-America, Africa, South-East Asia
* 18-70 years
* traveling for 1-10 weeks

Exclusion Criteria:

* Chronic diarrhea
* Pregnant
* Colitis Ulcerosa
* Morbus Chrohn
* IBS
* Coeliakie
* Gastrointestinal malabsorption
* microscopic colitis
* diverticulitis
* immune deficiency
* use of antibiotics/corticosteroids 2 weeks before travelling

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Travelers to tropical destinations visiting the outpatient clinic for vaccinations in a tertiary care hospital.
Sampling Method: Non-Probability Sample
Enrollment: 131 (Actual)
Dates: Start 2010-03; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
postinfectious IBS symptoms (ROME III criteria) 1 year after travelers diarrhea episode | 1 year after traveling

CONTACTS AND LOCATIONS:
Overall Officials: Guy Boeckxstaens, M.D., Principal Investigator — Catholic University Leuven
Locations (1):
- University hospitals Leuven, Leuven, Vlaams-Brabant, Belgium

REFERENCES:
- [Derived] Wouters MM, Van Wanrooy S, Nguyen A, Dooley J, Aguilera-Lizarraga J, Van Brabant W, Garcia-Perez JE, Van Oudenhove L, Van Ranst M, Verhaegen J, Liston A, Boeckxstaens G. Psychological comorbidity increases the risk for postinfectious IBS partly by enhanced susceptibility to develop infectious gastroenteritis. Gut. 2016 Aug;65(8):1279-88. doi: 10.1136/gutjnl-2015-309460. Epub 2015 Jun 12. PMID 26071133